CLINICAL TRIAL: NCT01310166
Title: A 6-month Multicenter, Single-arm, Open-label Study to Investigate Changes in Biomarkers After Initiation of Treatment With 0.5 mg Fingolimod (FTY720) in Patients With Relapsing-remitting Multiple Sclerosis
Brief Title: Biomarker Study After Initiation of Treatment With Fingolimod (FTY720) in Patients With Relapsing-remitting Multiple Sclerosis
Acronym: Biobank
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CFTY720DDE01; 2010-022066-28 (EudraCT Number)
Record Dates: First submitted 2011-02-24; First posted 2011-03-08 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Relapsing-remitting Multiple Sclerosis
Keywords: Multiple sclerosis; RRMS; relapsing-remitting; fingolimod; biomarkers
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Fingolimod Hydrochloride

ARMS (1):
- Fingolimod (Experimental)
  Interventions: Drug: Fingolimod

INTERVENTIONS:
Drug: Fingolimod

SUMMARY:
The purpose of this study is to investigate which changes in immunological biomarkers under treatment with fingolimod in patients with relapsing-remitting multiple sclerosis can be detected.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with relapsing forms of MS defined by 2005 revised McDonald criteria
* Patients with Expanded Disability Status Scale (EDSS) score of 0-6.5

Exclusion Criteria:

* Patients with a manifestation of MS other than relapsing remitting MS
* Patients with a history of chronic disease of the immune system other than MS such as known immunodeficiency syndrome
* History or presence of malignancy in the last 5 years
* Diabetic patients with moderate or severe non-proliferative diabetic retinopathy or proliferative diabetic retinopathy and uncontrolled diabetic patients
* Diagnosis of macular edema during Screening Phase
* Patients with active systemic bacterial, viral or fungal infections
* Negative for varicella-zoster virus IgG antibodies at Screening
* Patients who have been treated with cladribine, cyclophosphamide or mitoxantrone at any time
* History of cardiovascular disorder
* Women of child-baring potential and inadequate contraception

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2011-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Cluster of Differentiation (CD)4+ naive T cells (C-C Chemokine Receptor Type 7+(CCR7+CD45RA+) | 6 Months
Change from baseline of CD8+ naïve T cells (CCR7+CD45RA+) | 6 months
Change from baseline of CD4+ central memory T cells (CCR7+CD45RA-) | 6 months
Change from baseline of CD8+ central memory T cells (CCR7+CD45RA-) | 6 months
Change from baseline of CD8+ effector memory T-cells (CCR7-CD45RA-) | 6 months

SECONDARY OUTCOMES:
Change from baseline of B-lymphocytes | 6 months
Change from baseline of monocytes | 6 months
Change from baseline of Natural Killer cells | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (55):
- Germany (55):
  - Novartis Investigative Site, Ostfildern, Baden-Wurttemberg
  - Novartis Investigative Site, Altenholz-Stift, Germany
  - Novartis Investigative Site, Andernach, Germany
  - Novartis Investigative Site, Celle, Germany
  - Novartis Investigative Site, Dortmund, Germany
  - Novartis Investigative Site, Göttingen, Germany
  - Novartis Investigative Site, Kastellaun, Germany
  - Novartis Investigative Site, Kiel, Germany
  - Novartis Investigative Site, Krefeld, Germany
  - Novartis Investigative Site, Leipzig, Germany
  - Novartis Investigative Site, Leverkusen, Germany
  - Novartis Investigative Site, Mönchengladbach, Germany
  - Novartis Investigative Site, Aalen
  - Novartis Investigative Site, Abensberg
  - Novartis Investigative Site, Alzenau in Unterfranken
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Bad Mergentheim
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Berg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Böblingen
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Erbach im Odenwald
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Fulda
  - Novartis Investigative Site, Grevenbroich
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hennigsdorf
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Klingenmünster
  - Novartis Investigative Site, Lappersdorf
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Leverkusen
  - Novartis Investigative Site, Merzig
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Neuburg am Inn
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Schwendi
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Singen
  - Novartis Investigative Site, Stade
  - Novartis Investigative Site, Stadtroda
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Troisdorf
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Unterhaching
  - Novartis Investigative Site, Wermsdorf
  - Novartis Investigative Site, Wolfenbüttel